CLINICAL TRIAL: NCT00349219
Title: An International Randomized Phase III Study of First-line Erlotinib Followed by Second-line Cisplatin + Gemcitabine Versus First-line Cisplatin + Gemcitabine Followed by Second-line Erlotinib in Advanced Non Small Cell Lung Cancer
Brief Title: TORCH: A Study of Tarceva or Chemotherapy for the Treatment of Advanced Non Small Cell Lung Cancer
Acronym: TORCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: San Giuseppe Moscati Hospital (Other); Princess Margaret Hospital, Canada (Other); University of Alberta (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TORCH; 2005-005968-90 (EudraCT Number)
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: first-line; second-line; targeted therapy
MeSH Terms: interventions — Erlotinib Hydrochloride; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): erlotinib followed at progression by gemcitabine and cisplatin
  Interventions: Drug: erlotinib; Drug: cisplatin; Drug: gemcitabine
- 2 (Active Comparator): cisplatin and gemcitabine chemotherapy for 6 cycles, followed at progression by erlotinib
  Interventions: Drug: cisplatin; Drug: gemcitabine; Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — erlotinib 150 mg taken orally daily until disease progression
  Other Names: Tarceva
  Arms: 1
Drug: cisplatin — cisplatin 80 mg/m2 IV day 1 every 3 weeks given in second-line therapy
  Arms: 1
Drug: gemcitabine — gemcitabine 1200 mg/m2 IV days 1 and 8 every 3 weeks, given in second-line
  Arms: 1
Drug: cisplatin — cisplatin 80 mg/m2 IV day 1 every 3 weeks for 6 cycles
  Arms: 2
Drug: gemcitabine — gemcitabine 1200 mg/m2 IV days 1 and 8 every 3 weeks for 6 cycles
  Arms: 2
Drug: erlotinib — erlotinib 150 mg orally taken daily as second line therapy (after disease progression on chemotherapy)
  Other Names: Tarceva
  Arms: 2

SUMMARY:
The purpose of this study is to compare first-line erlotinib followed at progression by second-line chemotherapy vs. first-line chemotherapy followed at progression by second-line erlotinib in the treatment of Advanced Non Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Chemotherapy for patients affected by advanced NSCLC has demonstrated only modest improvement in survival rates over best supportive care: the prognosis of patients remains poor and the side effects are considerable. Therefore, novel agents are urgently needed for this disease. One way to improve effectiveness of therapies is to use non-chemotherapeutic agents that act on biological targets and cause fewer systemic side effects. Erlotinib(Tarceva)is a biological therapy that in recent clinical trials has shown promise in first- and second-line treatment of advanced NSCLC.

In this trial, patients will be randomized to one of two treatment strategies:

- erlotinib taken by mouth daily; and, if disease progression occurs, to be followed by chemotherapy with cisplatin and gemcitabine at standard doses for 6 cycles

OR

- chemotherapy with cisplatin and gemcitabine given intravenously at standard doses for 6 cycles; and if disease progression occurs to be followed by erlotinib taken by mouth daily

The study is conducted with the partial support of Roche, S.p.A.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cytologically or histologically confirmed non-small cell lung cancer
* Metastatic (stage IV) or locally advanced (stage IIIB, with metastasis to supraclavicular nodes or with pleural effusion).
* Both patients at first diagnosis or those with disease recurrence after former surgery are eligible.
* At least one target or non-target lesion according to RECIST criteria
* Male or female > 18 years of age (Italy upper age limit 70 years)
* ECOG PS 0 or 1
* Life expectancy of > 3 months
* Neutrophils > 1,500 mm3, platelets > 100,000 mm3, and hemoglobin > 9 g/dL
* Bilirubin level either normal or < 1.5 x ULN
* AST (SGOT) and ALT (SGPT) < 2.5 x ULN (< 5 x ULN if liver metastasis are present)
* Serum creatinine < 1.5 x ULN
* Effective contraception for both, male and female patients if the risk of conception exists
* Signed written informed consent

Exclusion Criteria:

* Prior exposure to agents directed at the HER axis (e.g. gefitinib, cetuximab, trastuzumab).
* Prior chemotherapy or therapy with systemic anti-neoplastic therapy (e.g., monoclonal antibody therapy) for advanced disease. Prior surgery and/or localised irradiation is permitted. Prior neoadjuvant chemotherapy for operable disease or adjuvant chemotherapy is permitted if it did not contain gemcitabine and if at least 1 year elapsed from the end of chemotherapy and the date of relapse.
* Any unstable systemic disease (including active infections, significant cardiovascular disease or myocardial infarction within the previous year, any significant hepatic, renal or metabolic disease), metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of study medications or render the patient at high risk from treatment complications.
* Any other malignancies within past 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or surgically resected prostate cancer with normal PSA).
* Patients are excluded if they have brain metastasis or spinal cord compression that has not yet been definitively treated with surgery and/or radiation; previously diagnosed and treated CNS metastases or spinal cord compression without evidence of stable disease (clinically stable imaging) for at least 2 months will also cause patients to be excluded. Patients with asymptomatic CNS metastases and not requiring steroids to control symptoms can be included, even if on anti-seizure medications.
* HIV positive patients
* Any inflammatory changes of the surface of the eye at baseline
* Patients who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
* Nursing and/or pregnant females
* Known or suspected hypersensitivity to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2006-12; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
overall survival | one year
progression free rate of first-line treatment with erlotinib | after 9 weeks of treatment

SECONDARY OUTCOMES:
toxicity | every 3 weeks during treatment, and every 3 months thereafter
progression-free survival | one year
quality of life during the first-line therapy | every 3 weeks during first-line therapy
prognostic biologic indicators | end of study
resource utilization | every 6 weeks during first-line therapy
response rate | at 9 and 18 weeks from treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — S.G. Moscati Hospital, Avellino, Italy; Charles Butts, M.D., Principal Investigator — University of Alberta, Cross Cancer Institute, Edmonton, Alberta, Canada; Fortunato Ciardiello, M.D., Ph.D., Principal Investigator — Second University of Naples, Italy; Chair Medical Oncology; Ronald Feld, M.D., Principal Investigator — Princess Margaret Hospital, Divison of Medical Oncology, Toronto, Ontario, Canada; Ciro Gallo, M.D., Ph.D., Principal Investigator — Second University of Naples, Italy; Chair Medical Statistics; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples, Italy; Director Clinical Trials Unit
Locations (73):
- Canada (15):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency Vancouver Island, Victoria, British Columbia
  - Cancer Care Mannitoba, Winnipeg, Manitoba
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Hôpital Régional de Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Durham Regional Cancer Centre, Oshawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - McGill University Cancer Centre, Montreal
- Italy (58):
  - ASL Viterbo Ospedale, Belcolle, (vt)
  - Azienda Sanitaria S. Giuseppe Moscati, Monteforte Irpino, AV
  - Istituto Oncologico di Bari, U.O. di Oncologia Medica e Sperimentale, Bari, BA
  - Università di Chieti, Cattedra di Oncologia Medica, Chieti, CH
  - Humanitas Centro Catanese di Oncologia, Catania, CT
  - Ospedale di Gaeta, Gaeta, LT
  - Ospedale S. Vincenzo di Taormina, Taormina, ME
  - Policlinico Universitario P. Giaccone, Palermo, PA
  - Casa di Cura La Maddalena S.p.A., Dipartimento Oncologico, Palermo, PA
  - Azienda Ospedaliera V. Cervello, Palermo, PA
  - Azienda Ospedaliera S. Maria degli Angeli, Servizio di Oncologia, Pordenone, PN
  - Ospedale di Prato, Prato, PO
  - Ospedale Civile di Faenza, Divisione di Oncologia Medica, Faenza, RA
  - Istituto Regina Elena, Divisione di Oncologia Medica, Roma, Roma
  - Ospedale S. Luca, Vallo della Lucania, SA
  - Ospedale San Lazzaro, Alba
  - Ospedale Cardinal Massaia, Asti
  - C.R.O. Istituto Nazionale Tumori, Aviano
  - Azienda Ospedaliera G. Rummo, Unità Operativa di Oncologia Medica, Benevento
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Ospedale A. Cardarelli, divisione Medicina Interna, Campobasso
  - Ospedale Ramazzini, Day Hospital Oncologico, Carpi
  - A.O. Ospedale Mater Domini, Oncoematologia Università Magna Grecia, Catanzaro
  - Ospedale Mariano Santo, U.O. di Oncologia Medica, Cosenza
  - Ospedale S. Corce, Fano
  - Azienda Ospedaliera Careggi, Florence
  - Azienda Ospedaliera Morgagni Pierantoni, Forlì
  - Ospedale Umberto I, U.O. di Oncologia Medica, Frosinone
  - Ospedale S. Martino, Genova
  - Ospedale Villa Scassi, Genova
  - Ospedale S. Maria Goretti, Latina
  - A.O. Vito Fazzi, Lecce
  - Ospedale C. Poma, Mantova
  - Policlinico Universitario G. Martino, Messina
  - Casa di Cura IGEA, Milan
  - Niguarda Ca' Granda, Milan
  - Ospedale L. Sacco, GISCAD Oncologia, Polo Universitario, Milan
  - Buon Consiglio Fatebenefratelli, Napoli
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Ospedale Cardarelli, Napoli
  - Second University of Naples, Napoli
  - Università Federico II, Cattedra di Oncologia Medica, Napoli
  - Divisione di Oncologia Medica, U.S.L.L. 13, Noale
  - Ospedale Civile Umbero I, Nocera Inferiore
  - Ospedale Civile di Nola, Reparto di Oncologia, Nola
  - Istituto Oncologico Veneto, Padua
  - Fondazione Salvatore Maugeri, Pavia
  - Ospedale S. Salvatore, Pesaro
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Azienda Ospedaliera S. Carol, Potenza
  - Ospedale degli Infermi, U.O. Oncologia Medica, Rimini
  - Ospedale S. Giovanni Calibita Fatebenefratelli, UO di Oncologia, Roma
  - Azienda Ospedaliera Universitaria Arcispedal, U.O. di Oncologia Clinica, Sant'Anna Di Ferrara
  - Azienda Ospedaliera Di Busto Arsizio, Saronno
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Ospedale E. Morelli, Sondalo
  - Azienda Sanitaria Locale 14, Verbania
  - Ospedale S. Andrea, Vercelli

REFERENCES:
- [Result] Gridelli C, Ciardiello F, Gallo C, Feld R, Butts C, Gebbia V, Maione P, Morgillo F, Genestreti G, Favaretto A, Leighl N, Wierzbicki R, Cinieri S, Alam Y, Siena S, Tortora G, Felletti R, Riccardi F, Mancuso G, Rossi A, Cantile F, Tsao MS, Saieg M, da Cunha Santos G, Piccirillo MC, Di Maio M, Morabito A, Perrone F. First-line erlotinib followed by second-line cisplatin-gemcitabine chemotherapy in advanced non-small-cell lung cancer: the TORCH randomized trial. J Clin Oncol. 2012 Aug 20;30(24):3002-11. doi: 10.1200/JCO.2011.41.2056. Epub 2012 Jul 9. PMID 22778317
- [Result] Di Maio M, Leighl NB, Gallo C, Feld R, Ciardiello F, Butts C, Maione P, Gebbia V, Morgillo F, Wierzbicki R, Favaretto A, Alam Y, Cinieri S, Siena S, Bianco R, Riccardi F, Spatafora M, Ravaioli A, Felletti R, Fregoni V, Genestreti G, Rossi A, Mancuso G, Fasano M, Morabito A, Tsao MS, Signoriello S, Perrone F, Gridelli C. Quality of life analysis of TORCH, a randomized trial testing first-line erlotinib followed by second-line cisplatin/gemcitabine chemotherapy in advanced non-small-cell lung cancer. J Thorac Oncol. 2012 Dec;7(12):1830-1844. doi: 10.1097/JTO.0b013e318275b327. PMID 23154555
- [Derived] Di Maio M, Gallo C, Leighl NB, Piccirillo MC, Daniele G, Nuzzo F, Gridelli C, Gebbia V, Ciardiello F, De Placido S, Ceribelli A, Favaretto AG, de Matteis A, Feld R, Butts C, Bryce J, Signoriello S, Morabito A, Rocco G, Perrone F. Symptomatic toxicities experienced during anticancer treatment: agreement between patient and physician reporting in three randomized trials. J Clin Oncol. 2015 Mar 10;33(8):910-5. doi: 10.1200/JCO.2014.57.9334. Epub 2015 Jan 26. PMID 25624439